CLINICAL TRIAL: NCT04835298
Title: Characters) Dyspnea Assessment in Adult Patients With Myotonic Dystrophy Type 1: a Monocentric Pilot Study
Brief Title: Breathlessness Assessment in Adult Patients With Myotonic Dystrophy Type 1
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20065*
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myotonic dystrophy type 1: adult patients with myotonic dystrophy type 1
  Interventions: Other: Dyspnea

INTERVENTIONS:
Other: Dyspnea — questionnaires

SUMMARY:
Myotonic dystrophy type 1 (DM1) is one of the most common neuromuscular diseases in adults. As respiratory dysfunction is the most common cause of death in patients with DM1, a respiratory disease progression must be monitored combining symptom screening and respiratory function testing, in order to identify the appropriate time to initiate non invasive ventilation (NIV).

Dyspnea, one of the main respiratory symptoms, has been little studied in patients with DM1.

The main objective of this study is to provide the first multidimensional description of dyspnea in patients with DM1.

The secondary objectives are:

* To compare respiratory symptoms according to the presence or not of criteria from respiratory function testing to initiate NIV
* To assess associations between dyspnea and respiratory function testing
* To assess associations between dyspnea and number of Cytosine Thymine Guanine (CTG) repeats
* To assess associations between dyspnea and muscular strength
* To assess associations between dyspnea and BMI
* To assess associations between dyspnea and anxiety or depression
* To assess associations between dyspnea and cognitive impairment
* To assess associations between dyspnea and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patient with myotonic dystrophy type 1 confirmed by genetic analysis
* with an age older than 18 years

Exclusion Criteria:

* an ongoing or recent (i.e. within the last 4 weeks prior to study recruitment) medical condition, including pulmonary exacerbations
* patient already under non-invasive mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with myotonic dystrophy type 1
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Dyspnea | Month 6
  Borg scale at rest and after 6 minute walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided